CLINICAL TRIAL: NCT07113054
Title: A Clinical Trial to Evaluate the Effect of Grapefruit Juice on the Pharmacokinetics and Pharmacodynamics of Edoxaban in Healthy Adults
Brief Title: A Clinical Trial to Evaluate the Effect of Grapefruit Juice on the PK/PD of Edoxaban
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hyewon Chung (Other)
Responsible Party: Sponsor-Investigator, Hyewon Chung, Assistant Professor, Korea University Guro Hospital
Organization: Korea University Guro Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EG-DDI
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Grapefruit Juice; Edoxaban
MeSH Terms: interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Edoxaban and Grapefruit Juice (Experimental): * Period 1: Single dose of edoxaban 60 mg administered alone
  * Period 2: Single dose of edoxaban 60 mg coadministered with grapefruit juice 3 times daily for 3 days
  Interventions: Drug: Edoxaban 60 MG [Lixiana]; Other: Edoxaban 60 MG [Lixiana] + Grapefruit Juice

INTERVENTIONS:
Drug: Edoxaban 60 MG [Lixiana] — Single administration of edoxaban
Other: Edoxaban 60 MG [Lixiana] + Grapefruit Juice — Coadministration of edoxaban and grapefruit juice

SUMMARY:
The aim of the study is to evaluate the effect of grapefruit juice on the pharmacokinetics and pharmacodynamics of edoxaban in healthy adults

DETAILED DESCRIPTION:
Pharmacokinetics and pharmacodynamics of edoxaban without coadministration of grapefruit juice will be compared with those after administration of grapefruit juice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 50 years of age (inclusive) at the time of screening
* Subjects with BMI of 18 to 32 kg/m2 (inclusive)
* Subjects who agree to use medically acceptable methods of contraception and not to donate sperm or oocyte
* Subjects who voluntarily decided to participate in the study and provided written consent to comply with the protocol

Exclusion Criteria:

* Subjects with current or history of clinically significant cardiovascular, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunological, dermatological, or neuropsychiatric disease
* Subjects with current or history of clinically significant hypersensitivity reactions or hypersensitivity reactions to the components or constituents of the investigational product
* Subjects who have clinically significant hemorrhage or increased risk of hemorrhage due to the following conditions A. Recent history of gastrointesinal ulcers B. Malignant tumor with a high risk of bleeding C. Recent brain or spinal cord injury D. Recent brain, spinal cord, or opthalmic surgery E. Recent history of intracranial or intracerebral hemorrhage F. Esophageal varices, arterial malformations, vascular aneurysms, or spinal cord or cerebral vascular abnormalities G. Coagulation disorders, thrombocytopenia, or platelet dysfunction H. Recent biopsy or major trauma I. Bacterial endocarditis J. Esophagitis, Gastritis, or Gastroesophageal reflux
* Subjects with a history of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Subjects whose eGFR calculated by the CKD-EPI formula is 80mL/min or less at Screening
* Subjects whose AST or ALT levels are more than 2 times the upper limit of normal range, or total bilirubin levels are more than 1.5 times the upper limit of normal range at screening
* Subjects whose coagulation test (aPTT, PT) exceeds the normal range at screening
* Subjects who have taken the following medication or medication known to have significant drug interactions with the investigational product within the 2 weeks prior to the first administration day A. Strong P-gp inhibitor or inducer B. Acetylsalicylic acid, antiplatelet agent, anticoagulant, fibrinolytic agent, non-steroidal anti-inflammatory drug (NSAID), selective serotonin reuptake inhibitor (SSRI), or selective serotonin-norepinephrine reuptake inhibitor (SNRI)
* Subjects who donated whole blood within 60 days or blood components within 30 days, or received blood transfusion within 30 days prior to the first administration day
* Subjects who participated and have been exposed to an investigational product in other clinical study within 180 days prior to the first administration day
* Subjects who consistently consumed alcohol (alcohol 21 units/week [1 unit = 10 g of pure alcohol]) within 2 weeks of the first administration day
* Subjects who consumed grapefruit or grapefruit juice within 2 weeks of the first administration day
* Pregnant or breastfeeding women
* Subjects judged unsuitable to participate in the clinical study by investigators due to other reasons, including the results of laboratory tests

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Cmax | 24 hours post-dose
  maximum concentration
AUCinf | 24 hours post-dose
  Area under the concentration-time curve from time of administration extrapolated to infinity
PT | 24 hours post-dose
  prothrombin time
aPTT | 24 hours post-dose
  activated partial thromboplastin time
TGA | 24 hours post-dose
  Thrombin generation assay

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Mendell J, Zahir H, Matsushima N, Noveck R, Lee F, Chen S, Zhang G, Shi M. Drug-drug interaction studies of cardiovascular drugs involving P-glycoprotein, an efflux transporter, on the pharmacokinetics of edoxaban, an oral factor Xa inhibitor. Am J Cardiovasc Drugs. 2013 Oct;13(5):331-42. doi: 10.1007/s40256-013-0029-0. PMID 23784266
- [Background] Ogata K, Mendell-Harary J, Tachibana M, Masumoto H, Oguma T, Kojima M, Kunitada S. Clinical safety, tolerability, pharmacokinetics, and pharmacodynamics of the novel factor Xa inhibitor edoxaban in healthy volunteers. J Clin Pharmacol. 2010 Jul;50(7):743-53. doi: 10.1177/0091270009351883. Epub 2010 Jan 15. PMID 20081065
- [Background] Liu L, Li X, Liu Y, Xu B, Li Y, Yuan F, Zhang P, Tu S, Hu W. Bioequivalence and Pharmacokinetic Study of 2 Edoxaban Tablets in Healthy Chinese Subjects. Clin Pharmacol Drug Dev. 2022 Dec;11(12):1440-1446. doi: 10.1002/cpdd.1156. Epub 2022 Aug 11. PMID 35950601
- [Background] Wang EJ, Casciano CN, Clement RP, Johnson WW. Inhibition of P-glycoprotein transport function by grapefruit juice psoralen. Pharm Res. 2001 Apr;18(4):432-8. doi: 10.1023/a:1011089924099. PMID 11451028
- [Background] Mikkaichi T, Yoshigae Y, Masumoto H, Imaoka T, Rozehnal V, Fischer T, Okudaira N, Izumi T. Edoxaban transport via P-glycoprotein is a key factor for the drug's disposition. Drug Metab Dispos. 2014 Apr;42(4):520-8. doi: 10.1124/dmd.113.054866. Epub 2014 Jan 23. PMID 24459178